CLINICAL TRIAL: NCT04055818
Title: Proof-of-concept Study of Nicotinamide and Oral Tetrahydrouridine (THU) and Decitabine to Treat High Risk Sickle Cell Disease
Brief Title: A Study of Nicotinamide With Oral Tetrahydrouridine and Decitabine to Treat High Risk Sickle Cell Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: EpiDestiny, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0631
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Niacinamide; Decitabine; Tetrahydrouridine

STUDY DESIGN:
Intervention Model Description: 1:1 Randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nicotinamide (Experimental): Oral Nicotinamide 1000 mg twice daily
  Interventions: Drug: Nicotinamide
- THU Decitabine (Experimental): Oral 250 mg THU and 5 mg decitabine Once per week
  Interventions: Drug: Nicotinamide

INTERVENTIONS:
Drug: Nicotinamide — Oral nicotinamide (Vitamin B3) alone compared to THU Decitabine combination
  Other Names: Decitabine; Tetrahydrouridine

SUMMARY:
A randomized control trial in 20 subjects with sickle cell disease comparing oral THU-decitabine to nicotinamide and in combination (THU, decitabine and nicotinamide).

DETAILED DESCRIPTION:
A randomized control trial comparing oral THU-decitabine to nicotinamide (1:1 randomization), and then comparing the effects of the combination of nicotinamide with THU-decitabine vs either treatment alone. Treatment with each agent alone is for 12 weeks followed by the combination for a further 12 weeks. Patients have the option to enter an extension phase of combination treatment for an additional 24 weeks (total of 48 weeks)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Written informed consent provided by the subject before study entry.
* Confirmed sickle cell disease (SCD) as determined by hemoglobin electrophoresis or liquid chromatography.
* Subject is in his/her steady state and not having any acute complication due to SCD (i.e., hospitalization, acute pain, or acute chest syndrome in the past 14 days).
* Weight at least 40kg
* Regular compliance with comprehensive care and previous therapy.
* Symptomatic SCD is defined as having one of following, despite at least 6 months of hydroxyurea therapy, or refuse to take hydroxyurea for personal reasons: fetal hemoglobin <0.5 g/dL, or 3 or more pain episodes per year requiring parenteral narcotics, or 1 or more acute chest syndrome episodes, or Hemoglobin <9 g/dL and absolute reticulocyte count <250,000/mm3.

Exclusion Criteria:

* Inability to give informed consent.
* Experienced severe sepsis or septic shock within the previous 12 weeks.
* Last HU dose was ingested within the previous 4 weeks.
* Currently pregnant or breast-feeding.
* Alanine Aminotransferase (ALT) ≥ 3 times the upper limit of normal or albumin <2.0 mg/dL or direct (conjugated) bilirubin ≥ 1.5 mg/dl.
* Serum creatinine >2.9 mg/dL and calculated creatinine clearance <30 mL/min.
* Platelet count >800 x 109/L.
* Absolute neutrophil count <1.5 x 109/L.
* Female of active childbearing potential who is unwilling to use at least one of the two following forms of birth control: (i) not having heterosexual sexual contact beginning at the screening visit and continuing until 4 weeks after the last dose of decitabine OR (ii) intrauterine device (IUD).
* Sexually active male who is unwilling to use a condom when engaging in any sexual contact with a female with child-bearing potential, beginning at the screening visit and continuing until 4 weeks after taking the last dose of THU and decitabine. This requirement applies also to males who have had a successful vasectomy.
* Altered mental status or recurrent seizures requiring anti-seizure medications.
* Moribund or any concurrent disease (e.g., hepatic, renal, cardiac, metabolic) of such severity that death within 24 weeks is likely.
* Concurrent diagnosis of malignancy including known Myelodysplastic syndrome, leukemia, or an abnormal karyotype.
* New York Heart Association (NYHA) class III/IV status.
* Eastern Co-operative Oncology Group (ECOG) performance status ≥3.
* Participant is on chronic transfusion therapy
* Known history of illicit drug or alcohol abuse within the past 12 months.
* Other experimental or investigational drug therapy in the past 28 days.
* Taking l-glutamine within the last 28 days
* Being positive for HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-24 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Blood Hemoglobin | 12 weeks
  Measure hemoglobin function

CONTACTS AND LOCATIONS:
Overall Officials: Robert Molokie, Principal Investigator — University of Illinois at Chicago College of Medicine
Locations (1):
- University of Illinois at Chicago College of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No